CLINICAL TRIAL: NCT03449563
Title: Effects of Open Thoracic Paravertebral Block on Postoperative Analgesia in Patients Undergoing Open Pulmonary Lobectomy
Brief Title: Effects of Open Thoracic Paravertebral Block on Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Wenya Bai, Resident dictor, Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nerve block
Record Dates: First submitted 2018-02-11; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: thoracic paravertebral block; postoperative analgesia; pulmonary lobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Placebo group (group G) (Placebo Comparator)
  Interventions: Other: placebo
- Ultrasound-guided TPVB group (group U) (Active Comparator)
  Interventions: Combination Product: Ultrasound-guided TPVB
- open TPVB group(group E) (Experimental)
  Interventions: Combination Product: Open TPVB

INTERVENTIONS:
Combination Product: Open TPVB — In Group E,the thoracic paravertebral block was performed under the direct vision with 0.25% ropivacaine 30 ml,and the Patient-controlled intravenous analgesia was administer after the surgery.
  Arms: open TPVB group(group E)
Combination Product: Ultrasound-guided TPVB — In Group U, thoracic paravertebral block was performed on the operated side under ultrasound guidance with 0.25% ropivacaine 30 ml,and the Patient-controlled intravenous analgesia was administer after the surgery.
  Arms: Ultrasound-guided TPVB group (group U)
Other: placebo — In Group G,patients were just received Patient-controlled intravenous analgesia after the surgery.
  Arms: Placebo group (group G)

SUMMARY:
The study was aimed to assess the effects of open thoracic paravertebral block on postoperative analgesia in patients undergoing open pulmonary lobectomy under general anesthesia. Then, A total of 90 patients with American Society of Anesthesiologists (ASA) scores of Ⅰ or Ⅱ, scheduled for open pulmonary lobectomy under propofol - remifentanil total intravenous anaesthesia, were randomly divided into PCIA group (group G), Ultrasound-guided TPVB combined with PCIA group (group U), and open TPVB combined with PCIA group (group E).Finally, the study find that Open TPVB can provided satisfactory analgesia for patients undergoing open pulmonary lobectomy under general anesthesia, and the analgesia efficacy was equivalent to the TPVB under ultrasound guidance,which should be popularized.

DETAILED DESCRIPTION:
Purpose: The study was aimed to assess the effects of open thoracic paravertebral block on postoperative analgesia in patients undergoing open pulmonary lobectomy under general anesthesia.

Methods: A total of 90 patients with American Society of Anesthesiologists (ASA) scores of Ⅰ or Ⅱ, scheduled for open pulmonary lobectomy under propofol - remifentanil total intravenous anaesthesia, were randomly divided into 3 groups (n = 30 each) by using a random number table: PCIA group (group G), Ultrasound-guided TPVB combined with PCIA group (group U), and open TPVB combined with PCIA group (group E). In group G, patients were received PCIA after the surgery. In group U, TPVB was performed on the operated side under ultrasound guidance with 0.25% ropivacaine 30 ml combined with the PCIA after the surgery. In group E, the TPVB was performed under the direct vision with 0.25% ropivacaine 30 ml combined with the PCIA. The Visual Analogue Score (VAS) at rest and during coughing, the sensory nerve block segment, as well as the respiratory rate were measured and recorded at different time-points. Furthermore, the hemodynamic vital signs at different time - points, the number of successfully delivered doses 48 h after the surgery, as well as the incidence of postoperative complications were also recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* with American Society of Anesthesiologists physical status Ⅰor Ⅱ
* aged 35 - 75 years old
* with body mass index of 20 - 25 kg／m2,
* scheduled for open pulmonary lobectomy under general anaesthesia at the First Affiliated Hospital of Kunming Medical University

Exclusion Criteria:

* cardiovascular and/or cerebrovascular disease;
* diabetes; pre-existing liver, lung or kidney dysfunction;
* bilateral surgery; take operations again within 48 h after the surgery;
* with serious pulmonary infection and coagulation dysfunction

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Score at rest | 30 minutes after extubation,1 hour after extubation, 2 hour after extubation, 4 hour after extubation, 6 hour after extubation, 8 hour after extubation, 12 hour after extubation, 24 hour after extubation, 48 hour after extubation
  Visual Analogue Score at rest was recorded at 30 minutes after extubation,1 hour after extubation, 2 hour after extubation, 4 hour after extubation, 6 hour after extubation, 8 hour after extubation, 12 hour after extubation, 24 hour after extubation, 48 hour after extubation. And the Visual Analogue Score was ranged from 0 to 10 (0 = no pain and 10 = worst pain imaginable).
Change in Visual Analogue Score during coughing | 30 minutes after extubation,1 hour after extubation, 2 hour after extubation, 4 hour after extubation, 6 hour after extubation, 8 hour after extubation, 12 hour after extubation, 24 hour after extubation, 48 hour after extubation
  Visual Analogue Score (VAS) during coughing was recorded 30 minutes after extubation,1 hour after extubation, 2 hour after extubation, 4 hour after extubation, 6 hour after extubation, 8 hour after extubation, 12 hour after extubation, 24 hour after extubation, 48 hour after extubation. And the Visual Analogue Score was ranged from 0 to 10 (0 = no pain and 10 = worst pain imaginable).
Change in the respiratory rate | 30 minutes after extubation,1 hour after extubation, 2 hour after extubation, 4 hour after extubation, 6 hour after extubation, 8 hour after extubation, 12 hour after extubation, 24 hour after extubation, 48 hour after extubation.
  The respiratory rate was recorded at 30 minutes after extubation,1 hour after extubation, 2 hour after extubation, 4 hour after extubation, 6 hour after extubation, 8 hour after extubation, 12 hour after extubation, 24 hour after extubation, 48 hour after extubation.

SECONDARY OUTCOMES:
Change in Blood pressure | immediately after the nerve block, 5 minutes after the nerve block, 10 minutes after the nerve block, 15 minutes after the nerve block, 20 minutes after the nerve block, 30 minutes after the nerve block, 45 minutes after the nerve block, 1 hour after the
  The blood pressure was recorded at the time points of immediately after the nerve block, 5 minutes after the nerve block, 10 minutes after the nerve block, 15 minutes after the nerve block, 20 minutes after the nerve block, 30 minutes after the nerve block, 45 minutes after the nerve block, 1 hour after the nerve block, 2 hour after the nerve block.
Change in Heart Rate | immediately after the nerve block, 5 minutes after the nerve block, 10 minutes after the nerve block, 15 minutes after the nerve block, 20 minutes after the nerve block, 30 minutes after the nerve block, 45 minutes after the nerve block, 1 hour after the
  The Heart Rate was recorded at the time points of immediately after the nerve block, 5 minutes after the nerve block, 10 minutes after the nerve block, 15 minutes after the nerve block, 20 minutes after the nerve block, 30 minutes after the nerve block, 45 minutes after the nerve block, 1 hour after the nerve block, 2 hour after the nerve block.
Change in pulse oximetry | immediately after the nerve block, 5 minutes after the nerve block, 10 minutes after the nerve block, 15 minutes after the nerve block, 20 minutes after the nerve block, 30 minutes after the nerve block, 45 minutes after the nerve block, 1 hour after the
  The pulse oximetry was recorded at the time points of immediately after the nerve block, 5 minutes after the nerve block, 10 minutes after the nerve block, 15 minutes after the nerve block, 20 minutes after the nerve block, 30 minutes after the nerve block, 45 minutes after the nerve block, 1 hour after the nerve block, 2 hour after the nerve block.
The number of successfully delivered doses of the patient-controlled intravenous analgesia pump | 48 hour after the surgery
  The number of successfully delivered doses of the patient-controlled intravenous analgesia pump was recorded 48 hour after the surgery.
The operating time of thoracic paravertebral block | From onset the thoracic paravertebral block to 24 hour after the surgery
The degree of parents'satisfaction with analgesia | up to three days after the surgery
  The degree of parents'satisfaction with analgesia was recorded three days after the surgery.
The postoperative complications like agitation, respiratory depression, nausea, vomiting | up to three days after the surgery
  The postoperative complications like agitation, respiratory depression, nausea, vomiting were recorded three days after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Zhao, Principal Investigator — First Affiliated Hospital of Kunming Medical University